CLINICAL TRIAL: NCT00961441
Title: An Open-Label, Multicenter, Parallel-Group, Two-Arm Study Comparing the Pharmacokinetics of Keppra XR in Children (Aged 12 - 16 Years Old) With Epilepsy and in Adults (Aged 18 - 55 Years Old) With Epilepsy
Brief Title: Study Evaluating the Pharmacokinetics of Keppra Extended Release (XR) in Children and Adults With Epilepsy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB BIOSCIENCES, Inc. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N01340; 2014-004376-39 (EudraCT Number)
Record Dates: First submitted 2009-08-17; First posted 2009-08-19 (Estimated); Results first posted 2011-05-25 (Estimated); Last update posted 2015-08-06 (Estimated); Status verified 2015-07

CONDITIONS: Epilepsy
Keywords: Levetiracetam; Epilepsy; Children; Adults
MeSH Terms: conditions — Epilepsy | interventions — Levetiracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Children 12-16 years old (Experimental)
  Interventions: Drug: Keppra XR
- Adults 18-55 years old (Experimental)
  Interventions: Drug: Keppra XR

INTERVENTIONS:
Drug: Keppra XR — Keppra XR 500 mg tablets and Keppra XR 750 mg tablets
  Dosage: Keppra XR 1000-3000 mg/day taken once daily. Duration: 4-7 days
  Other Names: Levetiracetam XR

SUMMARY:
To study how the body absorbs, distributes, metabolises and eliminates Keppra XR in both children (12 to 16 years old) and adults (18 to 55 years old) with epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a diagnosis of epilepsy on up to three concomitant anti-epileptic drugs
* Subjects on levetiracetam immediate release (IR) can be enrolled if on a stable dose for 7 days

Exclusion Criteria:

* Subjects with a history of status epilepticus within 3 months of Visit 1
* Subject has difficult venous accessibility

Ages: 12 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2009-09; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (6):
- United States (6):
  - Mobile, Alabama
  - Phoenix, Arizona
  - Little Rock, Arkansas
  - Fairfield, Connecticut
  - Bethesda, Maryland
  - Dallas, Texas

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Intent-to-treat (ITT) population includes all enrolled patients who received at least one dose of study medication.Pharmacokinetic Per-Protocol (PK-PP) population is a subset of the ITT population, consisting of those patients who had no major protocol deviations affecting the pharmacokinetic parameters.
Pre-assignment Details: Participant Flow and Baseline characteristics refer to the Intention-to-treat (ITT) population.
Groups:
- Keppra XR in Children (12-16 Years Old); Keppra XR in Adults (18-55 Years Old): Drug: Keppra XR
  Keppra XR 500 mg tablets and Keppra XR 750 mg tablets
  Dosage: Keppra XR 1000-3000 mg/day taken once daily
  Duration: 4-7 days
Period: Overall Study
Arm/Group | Keppra XR in Children (12-16 Years Old) | Keppra XR in Adults (18-55 Years Old)
Started | 12 | 13
Pharmacokinetic (PK-PP) Population | 12 | 10 (Two subjects were excluded due to study medication noncompliance, one due to wrong dosing regimen.)
Completed | 12 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Keppra XR in Children (12-16 Years Old) | Keppra XR in Adults (18-55 Years Old) | Total
Number analyzed (Participants) | 12 | 13 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.88 (1.37) | 41.78 (9.21) | 28.87 (15.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 6 | 5 | 11
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 77.2 (24.1) | 82.5 (23.0) | 80.0 (23.2)
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 165.9 (8.8) | 169.3 (10.3) | 167.7 (9.6)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 27.62 (7.01) | 28.63 (7.14) | 28.14 (6.95)
Body Surface Area (BSA) [Mean (Standard Deviation); unit: m^2] | 1.87 (0.34) | 1.95 (0.32) | 1.91 (0.32)
Race [Number; unit: Participants]
  Black | 4 | 3 | 7
  Caucasian | 8 | 9 | 17
  Other / mixed | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Maximum Concentration at Steady State (Cmax) of Keppra XR Normalized by Dose and by Body Weight and Dose During up to 7 Days of Administration
Description: The Cmax is the maximum plasma concentration normalized by dose and by body weight and dose.
  Cmax normalized by 1000 mg dose was calculated as:
  Cmax/(mg dose taken/ 1000 mg Keppra XR).
  Cmax normalized by body weight and dose (1 mg Keppra XR/kg) was calculated as:
  Cmax/(bodyweight (kg)/ mg dose Keppra XR taken).
  Pharmacokonetic (PK) samples were taken predose and 1h, 2.5h, 4h, 6h and 10h after study medication at day 4, 5, 6 or 7 of Keppra XR administration.
Time Frame: 6 pharmacokinetic samples were taken pre-dose, 1, 2.5, 4, 6 and 10 hours after administration, at Day 4, 5, 6, or 7 of Keppra XR administration.
Population: Pharmacokinetic Per-Protocol (PK-PP) population
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Keppra XR in Children (12-16 Years Old) | Keppra XR in Adults (18-55 Years Old)
Number analyzed (Participants) | 12 | 10
µg/mL
  Dose norm. ( Keppra XR 1000mg) | 17.3 [14.3 to 21.0] | 14.9 [12.1 to 18.5]
  Dose and weight norm. ( Keppra XR 1 mg/kg) | 1.27 [1.12 to 1.44] | 1.24 [1.08 to 1.42]
Statistical Analysis 1: Comparison: Keppra XR in Children (12-16 Years Old) vs Keppra XR in Adults (18-55 Years Old); An ANOVA for log-transformed values has been used as the basis for calculation of point estimates and Confidence Intervals (CIs); Test type: Superiority or Other; ANOVA; Point estimates for the geometric means ratios children/adults for Cmax normalized by dose and body weight and 90% CIs have been calculated; Point estimate for ratio = 1.0271, 90% CI 2-sided [0.8817 to 1.1964]

2. Primary Outcome: Area Under the Plasma Concentration Curve Over a Dosing Interval of 24 Hours (AUCtau) of Keppra XR Normalized by Dose, and by Body Weight and Dose During up to 7 Days of Administration
Description: AUCtau normalized by 1000 mg dose was calculated as:
  AUCtau/(mg dose taken/ 1000 mg Keppra XR).
  AUCtau normalized by body weight and dose (1 mg Keppra XR/kg) was calculated as:
  AUCtau/(bodyweight (kg)/ mg dose Keppra XR taken).
  6 PK samples were taken pre-dose, 1, 2.5, 4, 6 and 10 hours after administration, at Day 4, 5, 6, or 7 of Keppra XR administration. At steady state, reached after 2 days of administration of Keppra XR, the concentrations at 24h postdose is equal to the predose concentration. The predose concentration was used as the 24h concentration to calculate AUCτau.
Time Frame: as for outcome 1
Population: Pharmacokinetic Per-Protocol (PK-PP) population
Measure: Geometric Mean (95% Confidence Interval); unit: µg*h/mL
Arm/Group | Keppra XR in Children (12-16 Years Old) | Keppra XR in Adults (18-55 Years Old)
Number analyzed (Participants) | 12 | 10
µg*h/mL
  Dose norm. (Keppra XR 1000mg) | 265 [214 to 327] | 236 [187 to 298]
  Dose and weight norm. (Keppra XR 1 mg/kg) | 19.4 [16.5 to 22.9] | 19.6 [16.4 to 23.5]
Statistical Analysis 1: Comparison: Keppra XR in Children (12-16 Years Old) vs Keppra XR in Adults (18-55 Years Old); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ANOVA; Point estimates for the geometric means ratios children/adults for AUCtau normalized by dose and body weight and 90% CIs have been calculated; Point estimate for ratio = 0.9914, 90% CI 2-sided [0.8110 to 1.2118]

3. Primary Outcome: Time of Maximum Plasma Concentration (Tmax) of Keppra XR During up to 7 Days of Administration
Description: The Tmax is the time corresponding to the maximum plasma concentration of Keppra XR. It was directly obtained from the observed concentration versus time curve. 6 pharmacokinetic samples were taken pre-dose, 1, 2.5, 4, 6 and 10 hours after administration, at Day 4, 5, 6, or 7 of Keppra XR administration.
Time Frame: as for outcome 1
Population: PK-PP population
Measure: Median (Full Range); unit: hours (h)
Arm/Group | Keppra XR in Children (12-16 Years Old) | Keppra XR in Adults (18-55 Years Old)
Number analyzed (Participants) | 12 | 10
hours (h) | 5.90 [2.50 to 6.07] | 5.93 [2.45 to 6.05]

4. Primary Outcome: Apparent Total Body Clearance (CL/F) of Keppra XR During up to 7 Days of Administration
Description: The Apparent Total Body Clearance (CL/F) was calculated as Dose/ AUCtau. 6 pharmacokinetic samples were taken pre-dose, 1, 2.5, 4, 6 and 10 hours after administration, at Day 4, 5, 6, or 7 of Keppra XR administration.
Time Frame: as for outcome 1
Population: PK-PP population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Keppra XR in Children (12-16 Years Old) | Keppra XR in Adults (18-55 Years Old)
Number analyzed (Participants) | 12 | 10
L/h | 3.78 (31.4) | 4.23 (41.8)

5. Secondary Outcome: Occurrence of Treatment-Emergent Adverse Events From Starting Study Drug Treatment (Day 1) to up to 14 Days
Description: An Adverse Event (AE) is any untoward medical occurrence in a subject or clinical investigation subject administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. Treatment emergent means that an AE has begun or got worse after start of Keppra XR administration.
Time Frame: From Starting Study Drug Treatment (Day 1) to up to 14 days
Population: Safety Set includes all subjects who took at least one dose of study medication. The Safety Set is identical to the Intention-to-treat (ITT) population in this study.
Measure: Number; unit: Count
Arm/Group | Keppra XR in Children (12-16 Years Old) | Keppra XR in Adults (18-55 Years Old)
Number analyzed (Participants) | 12 | 13
Count
  Total number of AEs | 7 | 11
  Patients with at least 1 AE | 3 | 3
  Patients with severe AEs | 0 | 1
  Patients with serious AEs | 0 | 0

ADVERSE EVENTS:
Time Frame: From Starting Study Drug Treatment (Day 1) to up to 14 days.
Description: Treatment-Emergent AEs were collected and refer to the Safety Set. Safety Set includes all subjects who took at least one dose of study medication. Treatment emergent means that an Adverse Event has begun or got worse after start of Keppra XR administration.
Arm/Group | Keppra XR in Children (12-16 Years Old) | Keppra XR in Adults (18-55 Years Old)
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/13
Other Adverse Events (participants affected / at risk) | 3/12 | 3/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Keppra XR in Children (12-16 Years Old) (N=12) | Keppra XR in Adults (18-55 Years Old) (N=13)
Somnolence (Nervous system disorders) | 1 (1) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (2)
Fatigue (General disorders) | 1 (1) | 0 (0)
Irritability (General disorders) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Abnormal behaviour (Psychiatric disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 days but <= 180 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.